CLINICAL TRIAL: NCT05043636
Title: Diabetic Neuropathy Screening Study 1.1 + Substudy 1.2-1.3-1.4
Acronym: DANES
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: H-10929796
Record Dates: First submitted 2021-07-02; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Neuropathies; Distal Peripheral Sensory Neuropathy; Diabetic Foot; Foot Deformities; Autonomic Neuropathy; CAN
Keywords: vagus; sudoscan; rolltemp; hearttrends; pinprick; monofilament; MNSI; DN4
MeSH Terms: conditions — Diabetic Neuropathies; Diabetic Foot; Foot Deformities | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biological material to a biobank for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vagus — Cardiovascular autonomic neuropathy (Vagus) both resting heart rate variability and cardiovascular reflex tests The examination consists of 4 measures, all aimed at measuring heart rate. Measurements are taken for 5 minutes rest, change of position from lying to standing position, during deep breathing and by Valsalva (by breathing in a mouthpiece with a 40 mmHg resistance).
Device: HeartsTrends — • Cardiovascular autonomic neuropathy (HeartTrends®) measurers 60-minutes heart rate variability via a chest belt electrode (a Holter monitor) and an external data acquisition device.
Device: Sudoscan — Peripheral small-fiber sympathetic function (Sudoscan), measuring sudomotor function by electrochemical skin conductance in hands and feet
Device: UllMeter — • Pressure pain sensitivity of the chest bone is recorded (with a device which has the size and shape as a pen)during rest as a measure for sympathetic autonomic activity of the brain (UllMeter®) (www.stressmeter.org)
Device: DPN-check — Nerve conduction velocity and amplitude of the Sural nerves by DPN-check
Device: Rolltemp — Cold and warm sense of foot and lower leg
Device: Dexcom G6 Device — Insertion of continuous glucose monitor ( The Dexcom G6 Device)
  After 10 days in the study the patient will return the glucose monitor and diary by prepaid mail.
  Glycemic variability and hypoglycemia duration will be calculated from CGM data. Glycemic variability will be assessed by standard deviation (SD) and Coefficient of Variance (CV). We define normo-glycemic range as sensor glucose between 4.0 and 10.0 mmol/L. Hypoglycemia will be defined in two ranges as SG ≤3.9 mmol/L or SG ≤3.0 mmol/L). An episode of hypoglycemia will be defined as at least 15 minutes with SG below 3.9 mmol/L or 3.0 mmol/L, respectively. CGM recordings with less than 72 hours of data will be excluded from analysis.

SUMMARY:
The overall objective of this project is to describe the prevalence of and risk factors to diabetic neuropathy in a representative cohort of diabetes patients and to investigate pathophysiological conditions in those patients with neuropathy.

This project will yield substantial new knowledge about the prevalence of diabetic neuropathy in type 1 and type 2 DM persons, new risk factors to neuropathy and the association to other diabetic complications. Findings related to the study may facilitate new treatment regimens prompting a better neuropathy treatment with reduced incidence of diabetic complications.

First patients at SDCC will be screened for diabetic neuropathy (Study 1.1) with an extended neuropathy screening program as an addition to the routine neuropathy screening at SDCC. 1000 patients with type 1 DM and 1000 patients with type 2 DM will be included.

This screening study is a prerequisite for the further study of study participants in substudies investigating associations between diabetic neuropathy and diabetic complications as described below.

Hypothesis:

Several patients with diabetes have undiagnosed neuropathy and associated diabetic complications. We hypothesize that diabetic neuropathy is underdiagnosed at SDCC and can be diagnosed with targeted screening with new and traditional measuring techniques. In addition, several patients may have complications related to neuropathy, including foot complications, and dysregulation of glucose metabolism

Aim:

This study consists of a screening study (study 1.1) and two substudies (1.2 and 1.3 ). Study 1.1 is a cross-sectional study describing the prevalence of diabetic neuropathy based on questionnaire data and objective measures as described below and associated diabetic complications including foot complications.

The primary aim is to explore the prevalence of diabatic neuropathy in patients with type 1 and type 2 DM at SDCC and secondarily to explore associations between diabetic neuropathy and complications, as described in the respective sections below.

The substudy 1.2 is an observational single center cohort study with the aim of investigating associations between neuropathy diagnosed with new devices for measurement of neuropathy and foot complications in patients with type 1 and type 2 diabetes.

The substudy 1.3 is an observational single center cohort study investigating the association between CAN and glycemic variability in patients with type 1 diabetes.

DETAILED DESCRIPTION:
Study 1.1 Diabetic Neuropathy Screening Study Objective The objective of this study is to investigate the prevalence of diabetic neuropathy at the outpatient clinic of SDCC and to investigate the association between diabetic neuropathy and diabetic complications.

Aims Primary aims

* To describe the prevalence of the following kinds of diabetic neuropathy in a representative subset of type 1 and type 2 DM persons at SDCC:
* peripheral neuropathy assessed by traditional screening tools
* peripheral neuropathy assessed by novel screening tools
* autonomic neuropathy assessed by novel point-of-care screening tools
* peripheral and autonomic neuropathy assessed by validated neuropathy questionnaires

Secondary aims

* To explore the association between:
* the above-mentioned forms of neuropathy and possible risk factors for neuropathy such as HbA1c, urine albumin-creatinine-ratio, incidences of severe hypoglycaemia and ketoacidosis, BMI, vitamin B12, levels of SpO2 and quantitative measures of diabetic neuropathy
* the above-mentioned forms of neuropathy questionnaire data on mental health and wellbeing

Tertiary aim

•Study participants will be followed-up in national patient registries for mortality and morbidity at approximately 5, 10 and 15 years after examination and association studies to study outcomes and future disease and cause of death will be made Study Design: A cross-sectional study describing the prevalence of diabetic neuropathy based on questionnaire data and objective measures and their association to prevalent diabetic complications including. The duration of inclusion of participants in the study is estimated to be 3 years.

Measures:

Baseline data: Medication status, DM status, diagnoses of other diseases, diabetic complications, height, weight, retinopathy status, body mass index (BMI), smoking status, alcohol status Data collection and examinations: detailed description on "Groups and Interventions" Blood sugar Will be measured by capillary blood glucose measures of finger prick blood sample

Questionnaires:

All questionnaires are validated and in Danish. Compass 31, Michigan Neuropathy Screening (MNSI), DN4, Patient Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM), The gastrointestinal symptom rating scale (GSRS), The World Health Organization- Five Well-Being Index (WHO-5), Participant Health Questionnaire (PHQ-9), Pedersen-Bjergaard questionnaire, Gold questionnaire and others, Brief Pain Inventory (BPI), IIEF, FSFIF, DistressScale

Recruitment Participants will be recruited at two SDCC outpatient clinics: at Niels Steensens vej 4, 2860 Gentofte, Denmark and Gentofte Hospitalsvej 1, st. tv., 2900 Hellerup, Denmark.

Ethical approval Before study initiation the study will be approved by the regional ethical committee and by the Danish data protection agency.

Guidelines from Danish data protection guidelines be followed throughout the process. All patient data will be stored and treated in accordance with regulation 2016/679 from the European parliament on the protection of natural patients with regard to the processing of personal data and on the free movement of such data, dated 27 April 2016(27), and the Danish amendment to regulation 2016/679(28).

Statistics The associations between determinants and outcome measures will be estimated by using complete-case regression models adjusting for relevant confounders including age, sex and diabetes duration. Logistic regression analyses will be used for binary outcomes. Linear regression analyses will be used for continuous outcomes. Outcome variables will be log-transformed using the natural logarithm to meet model assumptions of the distribution of the model residuals if necessary. Interactions between sex and all determinants will be investigated in all models to investigate possible sex interactions differences. A level of significance of 5% will be used.

Sample size estimation: as this is a prevalence study a power calculation is not possible. As the aim is to describe neuropathy prevalence in a representative sample of patients, the investigators aim to assessed 50% of the patient population at SDCC by consecutively examining all patients at their yearly status examination. The investigators aim to examine 2000 participants in total.

Analyses will be performed using SAS version 9.3(SAS Institute, Cary, NC).

Substudy 1.2 Diabetic neuropathy and foot complications Objective The overall objective of this study is to investigate the association between diabetic neuropathy diagnosed with established and novel measuring techniques and foot complications Aims Primary aim •To describe the association between neuropathy diagnosed by novel point-of-care screening tools and foot complications in age and gender matched type 1 and type 2 diabetes patients at SDCC.

Secondary aim

•To compare the prevalence of foot complications in participants with neuropathy diagnosed by novel point-of-care screening tools and traditional point-of-care screening tools, in age and gender matched type 1 and type 2 diabetes patients at SDCC.

Participants:

300 participants older than 39 years of age with type 1 or type 2 diabetes at SDCC will be included in this study. The participants included must be diagnosed with peripheral neuropathy in the screening study. 150 participants with neuropathy diagnosed with novel assessment methods will be age and gender matched with 150 participants with neuropathy diagnosed with traditional methods.

Measures Results from neuropathy examinations and questionnaires are already sampled in study 1.1 and will be incorporated in the study.

Routine foot examination, which include

* Examination for foot ulcers, infection, cellosites, nail deformities, edema,
* Assessment of Charcot foot, walk, footwear

Expanded foot examination, which include:

* Assessment for deformities (Hallux valgus, hallux rigidus, pes planus, pes cavus, low forefoot, hammertoes, valgus/varus hindfod. Wide-ranging forefoot)
* Examination of the foot length and with
* 2 clinical photos with iphone (loaded and unloaded to Sundhedsplatformen) for clinical documentation.
* Assessment of insoles.

Statistics The associations between determinants and outcome measures will be estimated by using complete-case regression models adjusting for relevant confounders including age, sex and diabetes duration. Logistic regression analyses will be used for binary outcomes. Linear regression analyses will be used for continuous outcomes. Outcome variables will be log-transformed using the natural logarithm to meet model assumptions of the distribution of the model residuals if necessary. Interactions between sex and all determinants will be investigated in all models to investigate possible sex interactions differences. A level of significance of 5% will be used.

Analyses will be performed using SAS version 9.3 (SAS Institute, Cary, NC). Sample size estimation: as this is an exploratory study with no prior similar studies performed a power calculation is not possible. The investigators assess that comparing 150 participants diagnosed with novel assessment methods with 150 age and gender matched participants with neuropathy diagnosed with traditional methods will be sufficient to investigate differences in foot complication prevalence between the groups.

Substudy 1.3 Cardiovascular autonomy neuropathy and glucose variability Objective The overall objective of this study is to investigate if patients with type 1 diabetes and CAN have a larger glucose variability compared to similar patients without CAN.

Primary aim

* To investigate differences in SD (standard deviation) in 30 participants with and participants without CAN Secondary aims
* To investigate differences in CV (Coefficient of Variation), time spent in hyperglycaemia, time spent in hypoglycaemia, CONGA, MAGE in participants with and without CAN.
* To investigate associations between continuous measures of CAN and indices of glucose variability

Tertiary aims

* To investigate the association between CAN and hypoglycaemic unawareness.
* To investigate the association between symptoms of CAN and glucose variability.

Study Design 30 participants with type 1 diabetes with CAN will be enrolled and compare with 30 age and sex matched type 1 diabetes participants without CAN.

If it is not possible to enroll enough study participants patients will be recruited by using data from electronic patient records at SDCC containing data on 600 type 2 patients screened for CAN between 2013-2014. Information about civil registration number, phone number, address, diagnosis of type 1 diabetes, age, gender and historic data on CAN on outpatients at Steno Diabetes Center Copenhagen is provided by the treatment-responsible doctor and passed on to the study investigator. This information is used for identifying possible participants and recruitment. First contact will be a letter containing the written participant information and the brochure: "The participants rights as a participant in biomedical research". In the letter, possible participants will be invited to the information meeting at Steno Diabetes Center Copenhagen. The letter contains telephone number and email for the project-responsible doctor. Non-responders will be followed up by a telephone contact approximately two weeks later.

Power calculation As mentioned the CAN diagnosis has be shown to trend toward a significant association to CV by Nyiraty et al (39). With reference to that study the investigators hypotie that a difference in SD of 0.2 mmol/L is detectable (and relevant) between CAN and non-CAN patient. In this study the standard deviation of SD was approximately 0.2 mmol/L. With 90% power and a two-sided significance level of 0.05 the sample size needed to detect the abovementioned difference is 23 in each group - 46 participant in total. Taking a drop-out ratio of 10% into account and given the inaccurate nature of this power calculation the sample size of the study will be 30 participants in each group.

The prevalence of CAN at SDCC is 15 %. Thus, a screening of approximately 200 participants is needed to obtain the target participant number. 60 participants in total.

Methods and measures Participants Type 1 diabetes participants will be recruited from the screening (study 1.1.)

Methods CAN will be assessed by Cardiovascular reflex tests and heart rate variability indices (Vagus™ device).

Glucose variability will be assessed by use of 10 days continuous glucose monitoring attached to the skin of the participant with the Dexcom G6 sensor, transmitter and receiver. Several glucose variability indices will be assessed e.g. CV, MAGE, CONGA, time spent in hypoglycaemia, time spent in hyperglycemia.

Hypoglycemia unawareness will be assessed by the Pedersen-Bjergaard, the Gold questionnaire and others.

Measures

* Cardiovascular autonomic neuropathy testing with Vagustm device both resting heart rate variability and cardiovascular reflex tests (20 minutes) (as described in study 1.1)
* Insertion of continuous glucose monitor ( The Dexcom G6 Device) (15 minutes)

Recruitment Participants for this study will be participants who have been screened in study 1.1.

Statistics The associations between determinants and outcome measures will be estimated by using regression models adjusting for relevant confounders including age, sex and diabetes duration. Logistic regression analyses will be used for binary outcomes. Linear regression analyses will be used for continuous outcomes. Outcome variables will be log-transformed using the natural logarithm to meet model assumptions of the distribution of the model residuals if necessary. Interactions between sex and all determinants will be investigated in all models to investigate possible sex interactions differences. Analyses will be performed using SAS version 9.3 (SAS Institute, Cary, NC).

ELIGIBILITY:
Inclusion Criteria Study 1.1 Diabetic Neuropathy Screening Study :

* The ability to give informed consent
* Male or female persons >18 years of age with a diagnosis of type 1 or type 2 DM (WHO criteria)

Exclusion Criteria Study 1.1 Diabetic Neuropathy Screening Study:

* Ongoing cancer treatment or other concurrent illness that will make the participant unable to attend the study on the discretion of the investigator
* Pregnant or breastfeeding persons
* Persons who, in the judgement of the investigator, may not be able to follow protocol
* Persons in active laser treatment for retinopathy, will be excluded from only Valsalva test (part of CAN measurements)
* Persons with atrial fibrillation, atrial flutter or pacemakers will not be subjected to CAN measurements.

Inclusion Criteria Substudy 1.2 Diabetic neuropathy and foot complications

* The ability to give informed consent
* Male or female participants >39 years of age with a diagnosis of type 1 or type 2 diabetes (WHO criteria)
* Peripheral neuropathy diagnosed by either:
* Biothesiometry above age-stratified threshold values (150 participants) and/or abolished sensation to monofilament (10g) or
* Sudoscan and/or DPNCheck values below age-stratified threshold values (150 participants)

Exclusion Criteria Substudy 1.2 Diabetic neuropathy and foot complications

* Ongoing cancer treatment or other concurrent illness that will make the patient unable to attend the study on the discretion of the investigator
* Pregnant or breastfeeding participants
* Participants who, in the judgement of the investigator, may not be able to follow the protocol
* Participants in active laser treatment for retinopathy, will be excluded from only Valsalva test (part of Vagus™ measurements)
* Participants with atrial fibrillation, atrial flutter or pacemakers will not be subjected to CAN measurements.
* Participants with toe or foot amputations

Inclusion Criteria Substudy 1.3 Cardiovascular autonomy neuropathy and glucose variability

* Participants with type 1 diabetes, recruited from the screening study
* Participants with 20-80 of age

Exclusion Criteria Substudy 1.3 Cardiovascular autonomy neuropathy and glucose variability

* Pregnancy
* Participants who, in the judgement of the investigator, is incapable to participate
* Participants using insulin pumps
* Participants in beta-blocker treatment
* Participants with acute infection
* Participants with thyroid disease
* Participants with alcohol abuse
* Participants in active laser treatment for retinopathy, will be excluded from only Valsalva test (part of Vagus™ measurements)
* Participants with atrial fibrillation, atrial flutter or pacemakers will not be subjected to CAN measurements.
* Ongoing cancer treatment or other concurrent illness that will make the patient unable to attend the study on the discretion of the investigator. Participants treated with tricyclic antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with type 1 and type 2 DM attending Diabetes Mellitus treatment at Steno Diabetes Center Copenhagen will be invited to participate in this study. The persons will be recruited by receiving a letter describing the study.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Peripheral Neuropathy assesed by DPN-check | 18.10.2019-31.12.2022
  Neuropathy assesed by DPN-check:
  Sural Nerve conduction velocity(m/s) of the Sural nerves by DPN-check.
Autonomic Neuropathy assesed by Sudoscan | 18.10.2019-31.12.2022
  Neuropathy assesed by Sudoscan:
  Peripheral small-fiber sympathetic function (Sudoscan), measuring sudomotor function by electrochemical skin conductance (µS) in feet
Peripheral Neuropathy assesed by Biothesiometer | 18.10.2019-31.12.2022
  Neuropathy assesed by Biothesiometer:
  Peripheral vibration sensation (volt)
Peripheral Neuropathy assesed by Roll-temp | 18.10.2019-31.12.2022
  Neuropathy assesed by Roll-temp:
  Cold and warm sense of foot and lower leg by
Peripheral Neuropathy assesed by Monofilament | 18.10.2019-31.12.2022
  Neuropathy assesed by Monofilament Light touch with 10 and 75 g monofilament
Peripheral Neuropathy assesed by Pinprick | 18.10.2019-31.12.2022
  Neuropathy assesed by Pinprick:
  Pain Sensation with a 40g needle
Cardivascular Autonomic Neuropathy assesed by Vagus | 18.10.2019-31.12.2022
  The examination consists of 4 measures, all aimed at measuring heart rate. Measurements are taken for 5 minutes rest, change of position from lying to standing position, during deep breathing and by Valsalva (by breathing in a mouthpiece with a 40 mmHg resistance).

SECONDARY OUTCOMES:
Peripheral Neuropathy assesed by DPN-check | 18.10.2019-31.12.2022
  Neuropathy assesed by DPN-check: Sensory nerve action potential (amplitude) of the Sural nerves by DPN-check.
Autonomic Neuropathy assesed by Sudoscan | 18.10.2019-31.12.2022
  Neuropathy assesed by Sudoscan:
  Peripheral small-fiber sympathetic function (Sudoscan), measuring sudomotor function by electrochemical skin conductance (µS) in hands.
Pressure pain sensitivity | 18.10.2019-31.12.2022
  Pressure pain sensitivity of the chest bone is recorded (with a device which has the size and shape as a pen)during rest as a measure for sympathetic autonomic activity of the brain (UllMeter®) (www.stressmeter.org) (15 min, including 10 min. of rest)
Oxygen Saturation in supine and standing position | 18.10.2019-31.12.2022
  Oxygen saturation in supine and standing position (1, 2, 3, 4, 5 min.) (oxygen level in percentage)
Blood pressure in supine and standing position | 18.10.2019-31.12.2022
  Blood pressure (mmHg) in supine and standing position (1, 2, 3, 4, 5 min)

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark